CLINICAL TRIAL: NCT04810507
Title: A Multi-center, Active Controlled, Randomized, Double-blinded, Parallel, Phase IV Study to Evaluate the Effect of Improving Glycemic Variability of Anagliptin Compared With Sitagliptin in Patients With Type 2 Diabetes Mellitus
Brief Title: MAGE of Anagliptin Compared With Sitagliptin With Type 2 Diabetes Mellitus
Acronym: ACACIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWP-GDL-404
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A Multi-center, Active controlled, Randomized, Double-blinded, Parallel Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anagliptin arm (Experimental): Anagliptin 100 mg twice a day
  Interventions: Drug: Anagliptin BID Treatment
- Sitagliptin 100mg (Active Comparator): Sitagliptin 100mg once a day
  Interventions: Drug: Anagliptin BID Treatment

INTERVENTIONS:
Drug: Anagliptin BID Treatment — Continuous Glucose Monitoring with Anagliptin 100mg BID or Sitagliptin 100mg QD treatment for 12 weeks
  Other Names: Sitagliptin QD Treatment

SUMMARY:
An exploratory study to evaluate the Effect of Improving Glycemic Variability of Anagliptin Compared with Sitagliptin in Patients with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
This clinical trial is an exploratory study, and does not calculate the subject number based on statistical assumptions, and enrolls 50 subjects per group and a total of 100 subjects are registered to evaluate the effect of improving blood glucose variability in type 2 patients with anagliptin 100 mg twice a day(BID) and sitagliptin 100 mg once a day(QD).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM
* Metformin monotherapy for more than 8 weeks and metformin ≥ 1000 mg daily for more than 8 weeks.
* 6.5% ≤HbA1c< 8.5%
* Agreed Therapeutic Lifestyle change during the study period
* Obtained Informed Consent Form

Exclusion Criteria:

* Type 1 diabetes mellitus,
* History of intestinal obstruction
* NYHA class III to IV congestive heart failure,
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 X upper limit of normal (ULN) or Total bilirubin > 3 X ULN
* Creatinine clearance (CrCl)* < 50 mL/min
* Thyroid-stimulating hormone (TSH) ≥ 1.5 X ULN
* Allergic history for Anagliptin 또는 sitagliptin
* Being pregnant or nursing or suspected of being pregnant, or
* History of participation in other clinical studies in the preceding 3 months.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Effect of Improving Glycemic Variability | 3 days after 12 weeks treatment
  Mean amplitude of glycemic excursion (MAGE)

SECONDARY OUTCOMES:
Average nighttime (18:00~07:59) blood glucose change after 12 weeks compared to baseline | after 12 weeks treatment
  after 12 weeks compared to baseline in the test group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Jaewan Park, Study Director — JWPharmaceuticals
Locations (1):
- Kangdong Sacred Heart Hospital, Seoul, South Korea